CLINICAL TRIAL: NCT03976232
Title: Efficacy of Trans Cranial Direct Current Stimulation (tDCS) Along With Craniosacral Therapy (CST) on Sleep Disturbances in Patients With Chronic Low Back Pain (CLBP)
Brief Title: Trans Cranial Direct Current Stimulation Along With Craniosacral Therapy on Sleep Disturbances in Patients With Chronic Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Maharishi Markendeswar University (Deemed to be University) (Other)
Responsible Party: Principal Investigator, Subhasish Chatterjee, Subhasish Chatterjee, Maharishi Markendeswar University (Deemed to be University)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IEC-1361
Record Dates: First submitted 2019-05-27; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Sleep Disturbance; Chronic Low-back Pain
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- tDCS-Group (Experimental): Participants of this arm will receive tDCS and Conventional therapy for 2 weeks.
  Interventions: Device: Trans cranial Direct Current Stimulation (tDCS)
- CST- Group (Experimental): Participants of this arm will receive CST and Conventional therapy for 2 weeks.
  Interventions: Other: Craniosacral therapy (CST)
- combination of tDCS and CST (Active Comparator): Participants of this arm will receive CST+ tDCS and Conventional therapy for 2 weeks.
  Interventions: Other: tDCS+ CST

INTERVENTIONS:
Device: Trans cranial Direct Current Stimulation (tDCS) — Active tDCS will be applied for 20 minutes with 2 mA intensity. Anode will be placed at left dorsolateral prefrontal cortex and cathode will be placed at the right cerebellar cortex.
  Arms: tDCS-Group
Other: Craniosacral therapy (CST) — Craniosacral therapy will be given to all the participants which includes release of all major diaphragm, frontal lift, parietal lift, occipital lift, CV4 and dural tube rocking.
  Arms: CST- Group
Other: tDCS+ CST — This group will receive tDCS along with CST
  Arms: combination of tDCS and CST

SUMMARY:
Sleep problems in patients with CLBP are a very common complication and is the most neglected part of the management. Though previous literature suggested that sleep problems need to be managed in patients with CLBP, no physical therapy or manual therapy techniques has been checked for their efficacy to manage the same. Therefore, there is a need to check the efficacy of various physical therapy and manual therapy techniques so that sleep problems associated with CLBP can be managed effectively by physical means. The main purpose of the study is to check the efficacy of tDCS and CST to improve sleep, pain and quality of life in patients with CLBP.

ELIGIBILITY:
Inclusion Criteria:

1. People with chronic low back pain (more than 3 months)
2. Both males and females.
3. 18-50 years
4. Able to follow verbal commands.

Exclusion Criteria:

1. Diagnosed with primary sleep disorders
2. Pregnancy
3. Taking any medication for a psychological disorder
4. Acute or subacute LBP
5. Diagnosed with any other systemic disorder.
6. Spinal tumour.
7. Radicular pain and nerve root compression.
8. Severe spinal stenosis, spondylolisthesis, fibromyalgia.
9. Unstable angina and other cardiovascular disorders.
10. Malignancy.
11. History of other systemic and inflammatory disease.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-06 (Estimated); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-02-02 (Estimated)

PRIMARY OUTCOMES:
Polysomnography | changes between baseline to 2 weeks and 6 weeks
  Polysomnographic parameters will be recorded.
Pittsburgh sleep quality Index scale. | changes between baseline to 2 weeks and 6 weeks
  Qualitative assessment of sleep will be recorded by this scale

SECONDARY OUTCOMES:
Modified Oswestry disability index | changes between baseline to 2 weeks and 6 weeks
  Chronic low back pain-related disability will be recorded
NPRS | changes between baseline to 2 weeks and 6 weeks
  Pain intensity will be recorded

IPD SHARING:
Plan to Share IPD: No